CLINICAL TRIAL: NCT04447014
Title: Natural History Study of Children and Adults With Adrenocortical Cancer
Brief Title: Natural History Study of Children and Adults With Adrenocortical Cancer (ACC)
Status: Terminated | Type: Observational
Why Stopped: To avoid the duplication of resources and effort associated with the PI switching branches.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 200110; 20-C-0110
Record Dates: First submitted 2020-06-24; First posted 2020-06-25 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Adrenocortical Carcinoma; Adrenocortical Cancer
Keywords: Clinical Outcome; Advice in the Management of Cancer; Patterns of Disease Progression; Response or Lack of Response to Therapeutic Interventions; Natural History
MeSH Terms: conditions — Adrenocortical Carcinoma; Adrenal Cortex Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort 1: Subjects with confirmed adrenocortical cancer (ACC)

SUMMARY:
Background:

Adrenocortical cancer (ACC) is a rare tumor. The prognosis is very poor for people with advanced stages of ACC. Some people may live with ACC for years; others live for just months. Treatment options for ACC often do not work well. Researchers want to study the clinical course of the disease. They want to understand how adrenocortical cancer appear on imaging scans, how they respond to therapies, and the best treatment for them.

Objective:

To gain a better understanding of adrenal cancer.

Eligibility:

People ages 2 and older with ACC who are enrolled in NCI protocol 19-C-0016

Design:

Participants will be screened with a review of their medical records, tumor scans, and cancer test results and reports.

Participants may have CT and other scans. For the scans, they will lie in a machine that takes pictures of the body. They may have blood tests. They may have a 24-hour urine collection. They may be asked to sign a new consent form for some of these tests.

Participants will complete paper or electronic surveys. The surveys will ask about the effects of cancer on their emotional, physical, and behavioral well-being.

Participants will receive recommendations about how to manage their issues and potential treatment options for their cancer.

Participants home physician will be contacted every 6 to 12 months to collect medical information such as test results and scans.

Participants may be asked to return to the NIH every 6 to 12 months for follow-up tests.

Participants will contact study staff if there are any changes in their tumor.

Participants will be followed on this study for life.

DETAILED DESCRIPTION:
Background:

* Adrenocortical carcinoma (ACC) is a rare tumor with an incidence of 1.5 to 2 per million people per year. It has a very poor prognosis with an overall 5-year mortality rate of 75-90% and an average survival from the time of diagnosis of 14.5 months. Approximately 10% of ACC cases are associated with a hereditary cancer predisposition syndrome.
* The treatment of choice for a localized primary or recurrent tumor is surgical resection. Patients with recurrent or metastatic disease are infrequently curable by surgery alone.
* As with most solid tumors, chemotherapy options have limited benefit, although platinumbased therapies have response rates of 25 to 30%. To date no targeted therapy has been shown to be of any value in this disease. The role of neoadjuvant and adjuvant therapies, including systemic chemotherapy and radiotherapy, remains poorly defined and has been reported to have only a modest or no therapeutic effect.
* The natural history of ACC can vary greatly with some patients surviving only months while others can live with disease for years. The basis for these differing clinical presentations is not known. While one cannot exclude an immune or other host component as responsible for the diverse clinical courses, it is also possible that there may be a genetic basis for this phenomenon.
* Patients with rare tumors seek expert advice in the management of their care. A natural history study would establish a more formal mechanism for such referrals, while allowing the systematic collection of epidemiologic, genomic, molecular data.

Objective:

-Characterize the natural history of adrenocortical cancer (ACC). Data will include patient demographics, clinical characteristics, patterns of disease progression, response or lack of response to therapeutic interventions, disease recurrence and overall survival.

Eligibility:

* Subjects with documented ACC
* Age greater than or equal to 2 years old.

Design:

* This protocol is a subprotocol to protocol 19C0016 Natural History and Biospecimen Accrual Study for Children and Adults with Rare Solid Tumors . After enrollment on the master protocol and undergoing evaluations detailed in the master protocol, patients will be enrolled on this subprotocol specific for ACC.
* Medical history will be collected from medical records and patients followed throughout the course of their illnesses, with particular attention to patterns of disease recurrence and progression, response to therapies, duration of responses and hormone production in patients with hormone production as a manifestation of their disease, and patient reported outcomes. Tumor growth rates will also be calculated throughout the course of the disease.

ELIGIBILITY:
* INCLUSION CRITIERIA:
* Subjects enrolled into NCI protocol 19C0016 Natural History and Biospecimen Acquisition Study for Children and Adults with Rare Solid Tumors
* Subjects with histologically or cytologically documented ACC.
* Age greater than or equal to 2 years old
* Ability of subject or parent/guardian to understand and the willingness to sign a written consent document.

EXCLUSION CRITIERIA:

None

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: primary clinical
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2020-06-25 (Actual); Primary Completion 2022-06-27 (Actual); Study Completion 2023-01-12 (Actual)

PRIMARY OUTCOMES:
Characterize the natural history of adrenocortical cancer (ACC). Data will include clinical presentation, patterns of disease progression, response or lack of response to therapeutic interventions, disease recurrence and overall survival | 10 years
  Characterize the natural history of adrenocortical cancer (ACC). Data will include clinical presentation, patterns of disease progression, response or lack of response to therapeutic interventions, disease recurrence and overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Jaydira Del Rivero, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2020-C-0110.html